CLINICAL TRIAL: NCT01815866
Title: Cough-Generated Aerosols of Nontuberculous Mycobacteria in Patients With Cystic Fibrosis
Brief Title: Cough-Generated Aerosols of NTM in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Children's Miracle Network (Other); UF Peds (Unknown)
Responsible Party: Sponsor
Other Study IDs: 484-2012
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
Keywords: Positive Nontuberculous Mycobacteria
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum cultures
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CF with culturable NTM: CF patients who produce culturable aerosols of NTM will receive the following test: pulmonary function test, collecting a sputum culture if possible, coughing for 5 minutes into a tube connected to a canister, hypertonic saline and albuterol will be given after the 5 minutes of coughing and then they would repeat with another 5 minutes of coughing. There can be a break inbetween the coughing if needed.
  Interventions: Procedure: CF with culturable NTM

INTERVENTIONS:
Procedure: CF with culturable NTM — CF patients who produce culturable aerosols of NTM will receive the following test: pulmonary function test, collecting a sputum culture if possible, coughing for 5 minutes into a tube connected to a canister, hypertonic saline and albuterol will be given after the 5 minutes of coughing and then they would repeat with another 5 minutes of coughing. There can be a break inbetween the coughing if needed.

SUMMARY:
Non-tuberculous mycobacteria (NTM) are opportunistic pathogens normally found in soil and water that are being cultured from Cystic Fibrosis (CF) airways at an increasing frequency. They have been demonstrated to cause clinically significant lung disease in some cases and the transmission of NTM, from person to person has been proposed. There are currently no standardized guidelines for isolation of those colonized or infected with NTM.

The investigators will measure particle droplet size from patients with CF who have positive sputum cultures for NTM with the hypothesis that they will be in a range that can spread infection.

DETAILED DESCRIPTION:
Patients with a positive NTM sputum culture will be asked to participate in the study. If they agree to participate they will sign an informed consent and will be scheduled to come to the University of Florida Clinical Research Center for the testing.

The test will consist of the following: pulmonary function test, collecting a sputum culture if possible, coughing for 5 minutes into a tube connected to a canister, hypertonic saline and albuterol will be given after the 5 minutes of coughing and then they would repeat with another 5 minutes of coughing. There can be a break inbetween the coughing if needed.

Patients maybe asked to come back a second time if they develop a different type of NTM or start treatment for NTM.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to age 8 years
* Confirmed Diagnosis of CF
* Sputum/Throat/Bronchoscopic culture positive for NTM within the last 12 months

Exclusion Criteria:

* Pregnancy
* Pneumothorax within the last 6 months
* Forced Expiratory Volume at one second <30% predicted
* Hemoptysis greater than 1 tablespoon within the last 7 days

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specialialty Clinics, Pulmonary
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The number of CF patients who produce culturable aerosols of NTM during coughing. | 6 weeks
  Patients with CF and a positive sputum or bronchoalveolar lavage (BAL) culture for NTM will cough into a chamber filled with culture plates that can measure droplet size. The investigators are looking for large droplets, that could land on surfaces and be a source for infection transmission, as well as fine droplets(5 microns or less)that are consistent with airborne transmission.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela M Schuler, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Research Center, Gainesville, Florida, United States